CLINICAL TRIAL: NCT02433652
Title: A Phase 1 Evaluation of the Safety and Protective Efficacy of a Single Dose of a Trivalent Live Attenuated Dengue Vaccine to Protect Against Infection With DENV-2
Brief Title: Evaluating the Safety and Protective Efficacy of a Single Dose of a Trivalent Live Attenuated Dengue Vaccine to Protect Against Infection With DENV-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 300
Record Dates: First submitted 2015-04-27; First posted 2015-05-05 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Dengue
Keywords: Dengue Vaccine
MeSH Terms: conditions — Dengue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trivalent dengue vaccine admixture + rDEN2Δ30-7169 (Experimental): Participants will receive the trivalent dengue vaccine admixture at Day 0 and the rDEN2Δ30-7169 vaccine at Day 180.
  Interventions: Biological: Recombinant live attenuated trivalent dengue vaccine; Biological: rDEN2Δ30-7169 vaccine
- Placebo + rDEN2Δ30-7169 (Experimental): Participants will receive a placebo vaccine at Day 0 and the rDEN2Δ30-7169 vaccine at Day 180.
  Interventions: Biological: Placebo; Biological: rDEN2Δ30-7169 vaccine

INTERVENTIONS:
Biological: Recombinant live attenuated trivalent dengue vaccine — Contains 10^3.3 plaque forming units (PFU)/mL of rDEN1Δ30, 10^3.3 PFU/mL of rDEN3Δ30/31-7164 and 10^3.3 PFU/mL of rDEN4Δ30. It is administered in 0.5 mL containing 10^3.0 PFU of each component.
  Arms: Trivalent dengue vaccine admixture + rDEN2Δ30-7169
Biological: Placebo
  Arms: Placebo + rDEN2Δ30-7169
Biological: rDEN2Δ30-7169 vaccine — Live recombinant attenuated DENV-2 candidate vaccine virus; will be administered at a dose of 10^3 PFU

SUMMARY:
Infection with dengue viruses is the leading cause of hospitalization and death in children in many tropical Asian countries, and the development of a dengue vaccine is a top health priority. This study will evaluate the ability of a single dose of a trivalent dengue vaccine to protect against infection with an attenuated candidate DENV-2 vaccine, administered 6 months after the trivalent dengue vaccine.

DETAILED DESCRIPTION:
There are 4 types of dengue virus (DENV-1, DENV-2, DENV-3, and DENV-4), each capable of causing dengue illness ranging from a mild illness to life-threatening disease. This study will evaluate a trivalent live attenuated dengue admixture vaccine that contains 3 different monovalent dengue vaccine candidates, representing 3 of the 4 dengue serotypes (DENV-1, DENV-3, and DENV-4). Study researchers will evaluate the safety and protective efficacy of a single dose of the trivalent dengue vaccine against viremia and rash induced by infection with an attenuated DENV-2 virus (rDEN2Δ30-7169), administered 6 months after the trivalent dengue vaccine.

This study will enroll healthy adults with no history of previous flavivirus infection. At Day 0 (study entry), participants will be randomly assigned to receive either the trivalent dengue vaccine admixture or placebo. On Day 180, all participants will receive the rDEN2Δ30-7169 vaccine. Study visits will occur on Days 4, 6, 8, 10, 12, 14, 16, 21, 28, 56, 90, 150, 180, 184, 186, 188, 190, 192, 194, 196, 201, 208, 236, 270, and 360. Visits will include physical examinations and blood collection. All participants will record their temperature 3 times a day for 16 days after each vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female between 18 and 50 years of age, inclusive
* Good general health as determined by physical examination, laboratory screening, and review of medical history
* Available for the duration of the study, approximately 26 weeks post-second vaccination
* Willingness to participate in the study as evidenced by signing the informed consent document
* Females Only: Female participants of childbearing potential willing to use effective contraception. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, abstinence (6 months or longer since last sexual encounter). All female participants will be considered having child-bearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria:

* Females Only: Currently pregnant, as determined by positive beta-human choriogonadotropin (HCG) test, or breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Screening laboratory values of Grade 1 or above for absolute neutrophil (ANC), alanine aminotransferase (ALT), and serum creatinine, as defined in this protocol
* Any condition that in the opinion of the investigator would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Any significant alcohol or drug abuse in the past 12 months that has caused medical, occupational, or family problems, as indicated by participant history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* HIV infection, by screening and confirmatory assays
* Hepatitis C virus (HCV) infection, by screening and confirmatory assays
* Hepatitis B virus (HBV), by HBV surface antigen (HBsAg) screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following vaccination. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days
* Receipt of a live vaccine within 28 days or a killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination
* Asplenia
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination
* History of serologic evidence of previous dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis virus, West Nile virus)
* Previous receipt of a flavivirus vaccine (licensed or experimental)
* Anticipated receipt of any investigational agent in the 28 days before or after vaccination
* Participant has definite plans to travel to a dengue endemic area during the study
* Refusal to allow storage of specimen for future research

Inclusion Criteria for Second Vaccine:

* Good general health as determined by physical examination and review of medical history
* Available for the duration of the study, approximately 26 weeks after the second dose
* Females Only: Female participants of childbearing potential willing to use effective contraception. Reliable methods of contraception include: hormonal birth control, condoms with spermicide, diaphragm with spermicide, surgical sterilization, intrauterine device, abstinence (6 months or longer since last sexual encounter). All female participants will be considered having child-bearing potential except for those with hysterectomy, tubal ligation, tubal coil (at least 3 months prior to vaccination), or post-menopausal status documented as at least 1 year since last menstrual period.

Exclusion Criteria for Second Vaccine:

* Anaphylaxis or angioedema following the first dose of vaccine
* Females only: Currently pregnant, as determined by positive beta-HCG test or breastfeeding
* Evidence of clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease by history, physical examination, and/or laboratory studies
* Behavioral, cognitive, psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand and cooperate with the requirements of the study protocol
* Any condition that in the opinion of the investigator would jeopardize the safety or rights of a participant to understand and cooperate with the requirements of the study protocol
* Any significant alcohol or drug abuse in the past 12 months that has caused medical, occupational, or family problems, as indicated by participant history
* History of a severe allergic reaction or anaphylaxis
* Severe asthma (emergency room visit or hospitalization within the last 6 months)
* HIV infection, by screening and confirmatory assays
* HCV infection, by screening and confirmatory assays
* HBV infection, by HBsAg screening
* Any known immunodeficiency syndrome
* Use of anticoagulant medications
* Use of corticosteroids (excluding topical or nasal) or immunosuppressive drugs within 28 days prior to or following inoculation. Immunosuppressive dose of corticosteroids is defined as greater than or equal to 10 mg prednisone equivalent per day for greater than or equal to 14 days.
* Receipt of a live vaccine within 28 days or killed vaccine within the 14 days prior to vaccination or anticipated receipt of any vaccine during the 28 days following vaccination
* Asplenia
* Receipt of blood products within the past 6 months, including transfusions or immunoglobulin or anticipated receipt of any blood products or immunoglobulin during the 28 days following vaccination
* Anticipated receipt of any other investigational agent in the 28 days before or after vaccination
* Participant has definite plans to travel to a dengue endemic area during the study
* Refusal to allow storage of specimens for future research

Other Treatment and Ongoing Exclusion Criteria:

The following criteria will be reviewed on Study Days 28 and 56 following each vaccination. If any become applicable during the study, the participant will not be included in further immunogenicity evaluations, as of the exclusionary visit. The participant will, however, be encouraged to remain in the study for safety evaluations for the duration of the study.

* Use of any investigational drug or investigational vaccine other than the study vaccine during the 28-day period post-vaccination
* Chronic administration (greater than or equal to 14 days) of steroids (defined as prednisone equivalent of greater than or equal to 10 mg per day), immunosuppressants, or any other immune-modifying drugs initiated during the 28-day period post-vaccination (topical and nasal steroids are allowed)
* Receipt of a licensed vaccine during the 28-day period post vaccination
* Receipt of immunoglobulins and/or any blood products during the 28-day period post-vaccination
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Frequency of trivalent dengue vaccine admixture and rDEN2Δ30-7169-related adverse events (AEs) | Measured through Day 360
  Classified by both severity and seriousness, through active and passive surveillance.
Dengue virus neutralizing antibody titers (measured through blood collection) | Measured through Day 360

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins School of Public Health; Kristen Pierce, MD, Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Center for Immunization Research (CIR), Johns Hopkins School of Public Health, Baltimore, Maryland
  - University of Vermont, Burlington, Vermont